CLINICAL TRIAL: NCT05716685
Title: Evaluation of Health Coaching to Empowering Hospitalised Chronic Heart Failure Patients
Brief Title: Health Coaching to Empowering Hospitalised Chronic Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: HCEP
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Education; Nursing
Keywords: Health coaching; Intervention; Chronic heart failure; Empowerment
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 19 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Health coaching — The intervention consisted of transferring the knowledge acquired on health coaching by the nurses of the cardiology unit to their care activity with CHF patients. To this end, all the nurses in the cardiology unit received two training packages: 1) five theoretical and practical sessions on health coaching competencies, emotional intelligence, communication and support for CHF patients in the hospital setting; and 2) training sessions 7 months after the first training package to reinforce the theoretical and practical knowledge acquired in health coaching. During this period, debriefing was carried out to provide feedback on the health coaching process with patients.

SUMMARY:
Aims: To evaluate the preliminary efficacy of Health Coaching in empowering hospitalised chronic heart failure patients.

Methods: pre-post quasi-experimental pilot study was carried out with 59 patients, allocated into the pre-intervention group (N=29) and post-intervention group (N=30) in a cardiology ward of a hospital. The intervention consisted of the knowledge traslation acquired on health coaching by the nurses of the cardiology unit to their care activity with CHF patients. The Patient empowerment in long-term conditions Questionnaire was used to measure heart failure patients: Attitude and sense of control; Shared and informed decision-making; and Information seeking and peer sharing, on two occasions: T1, pre-intervention, and T2, after completion of the intervention.

DETAILED DESCRIPTION:
Data collection:

Data collection was carried out by two members of the research team, who were not directly involved in the care of the patients, at two points in time: T1, pre-intervention, and T2, post-intervention. Two questionnaires were used for data collection:

1. Patient empowerment questionnaire for patients with chronic illness (Garcimartin et al. 2019): validated instrument in Spain with good psychometric properties, excellent Cronbach's alpha (>0.9) and moderate interclass correlation coefficient (0.47). It consists of 47 items and 3 dimensions: 1) Positive attitude and sense of control (21 items); 2) Shared and informed decision-making (13 items); and 3) Information seeking and sharing among peers (13 items). Response options for each item are scored on a 5-point Likert-type scale (1 strongly disagree and 5 strongly agree). The overall score for each patient ranges from 47 (worst empowerment) to 235 (best empowerment).
2. Questionnaire to collect sociodemographic and clinical variables: sex, age, educational level, marital status, employment status, hospital stay, Charlson index, 10-year survival, functional class (I-IV; according to NYHA), time of diagnosis and admissions in recent months.

Ethical considerations:

This study conformed to the principles set out in the Declaration of Helsinki and was approved by the centre's board and by the Research Ethics Committee (code 2019.066). Data custody complied with Organic Law 3/2018 on data protection (LOPDE). Informed consents were given to all participants. They were informed verbally and in writing about their free participation, the confidentiality and anonymity of the data and its use for scientific purposes. Nobody declined to participate or withdrew at any point of the study.

ELIGIBILITY:
Inclusion Criteria:

1) ≥18 years old; (2) at any stage of their disease (I-IV), according to the New York Heart Association Functional Class (NYHA) classification; (3) who had been admitted for more than 3 days; (4) whose level of consciousness was normal and whose state of health allowed them to complete the questionnaire; (5) who spoke and understood Spanish and; (6) who signed the informed consent form.

Exclusion Criteria: Patients with cognitive impairment or unable to answer the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Attitude and sense of control (21 items); Shared and informed decision-making (13 items); and Information seeking and peer sharing (13 items) | T1, pre-intervention ( 2019 August - 2020 February)
  Measurement tool: The Patient empowerment in long-term conditions Questionnaire
Attitude and sense of control (21 items); Shared and informed decision-making (13 items); and Information seeking and peer sharing (13 items) | T2, after completion of the intervention (2021 January - 2022 March) .
  Measurement tool: The Patient empowerment in long-term conditions Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Paloma, MD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- UCEC, Pamplona, Navarre, Spain

REFERENCES:
- [Result] Paloma B, Olano-Lizarraga M, Rumeu-Casares C, Quesada A, Saracibar-Razquin M, Vazquez-Calatayud M. [Level of empowerment of hospitalized chronic heart failure patient]. An Sist Sanit Navar. 2021 Dec 27;44(3):351-360. doi: 10.23938/ASSN.0960. Spanish. PMID 34142990
- [Result] Perez Paloma P, Gonzalez Urmeneta I, Roda-Casado C, Vazquez-Calatayud M. [A systematic review of interventions to empower patient with chronic heart failure in hospital environment]. An Sist Sanit Navar. 2020 Dec 22;43(3):393-403. doi: 10.23938/ASSN.0925. Spanish. PMID 33275128